CLINICAL TRIAL: NCT07250152
Title: Enhanced Prediction Model for Major Adverse Events Following Acute Myocardial Infarction
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1224
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction (MI)
Keywords: myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MI group: Patients who present with myocardial infarction and undergo successful percutaneous coronary intervention will be eligible for enrollment.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention

SUMMARY:
Acute myocardial infarction (AMI) remains a leading cause of mortality worldwide. Although early revascularization has markedly improved short-term outcomes, the incidence of major adverse cardiovascular events after the index event remains unacceptably high, posing a formidable clinical challenge. Contemporary risk-stratification instruments rely predominantly on a restricted set of conventional clinical variables and therefore fail to capture the full spectrum of individual pathophysiological complexity. To overcome these limitations, the present investigation aims to develop a post-AMI prognostic model that integrates comprehensive multimodal data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Presented with myocardial infarction, including NSTEMI and STEMI
3. Undergoing successful percutaneous coronary intervention.

Exclusion Criteria:

1. Subjects who decline protocol-mandated follow-up or withhold informed consent.
2. Individuals whose expected survival is < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myocardial infarction
Sampling Method: Probability Sample
Enrollment: 1544 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent myocardial infarction or cardiac death | At 24-month Follow-up
  Patients received recurrent myocardial infarction or cardiac death
Diagnostic performance | At 24-month follow-up
  Diagnostic performance of the AI-driven multimodal predictive model: area under the receiver-operating characteristic curve (AUC), sensitivity, specificity, overall accuracy, positive predictive value (PPV), and negative predictive value (NPV).
MACE at 24 months | At 24-month follow-up
  Major adverse cardiovascular events, defined as a compisite of cardiac death, myocardial infarction, target vessel revascularization.

SECONDARY OUTCOMES:
MACE at 60 months | At 60-month follow-up
  Major adverse cardiovascular events, defined as a compisite of cardiac death, myocardial infarction, target vessel revascularization.

OTHER OUTCOMES:
MACE according to pre-specified subgroups | At 24- and 60-month follow-up
  MACE stratified by sex, diabetes status, and chronic kidney disease (CKD) status.
MACE according to physiological status | At 24- and 60-month follow-up
  MACE prediction integrating physiological metrics-angiographic FFR, IMR, MRR, and CFR-of the culprit and non-culprit coronary arteries.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No